CLINICAL TRIAL: NCT02515669
Title: A Multi-Site, Randomized, Placebo-Controlled, Double-Blind, Multiple Ascending Subcutaneous Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of RO7239361 (BMS-986089) in Ambulatory Boys With Duchenne Muscular Dystrophy
Brief Title: Study of an Investigational Drug, RO7239361 (BMS-986089), in Ambulatory Boys With DMD
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: A pre-planned futility analysis indicated lack of efficacy in study NCT03039686 and led to discontinuation of both ongoing studies in DMD.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CN001-006; WN40226 (Other: Hoffman-La Roche)
Record Dates: First submitted 2015-07-29; First posted 2015-08-05 (Estimated); Results first posted 2019-05-08 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-10

CONDITIONS: Muscular Dystrophy (DMD)
MeSH Terms: conditions — Muscular Dystrophies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RO7239361 (Active Comparator): RO7239361 subcutaneous injections on specified days
  Interventions: Drug: RO7239361
- Placebo (Placebo Comparator): Placebo subcutaneous injections on specified days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RO7239361 — Colorless to slightly yellow, clear to opalescent solution, essentially free of particulate matter packaged in a 1 cc glass syringe equipped with a safety syringe device.
  Other Names: Anti-Myostatin Adnectin; taldefgrobep alfa
  Arms: RO7239361
Drug: Placebo — Colorless to slightly yellow, clear to opalescent solution, essentially free of particulate matter packaged in a 1 cc glass syringe equipped with a safety syringe device.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety and tolerability of RO7239361 in boys with Duchenne Muscular Dystrophy with any genetic mutation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with DMD
* Able to walk without assistance
* Able to walk up 4 stairs in 8 seconds or less
* Weigh at least 15 kg
* Taking corticosteroids for DMD

Exclusion Criteria:

* Ejection fraction < 55% on echocardiogram, based on central read
* Any behavior or mental issue that will affect the ability to complete the required study procedures
* Previously or currently taking medications like androgens or human growth hormone
* Use of a ventilator during the day
* Unable to have blood samples collected or receive an injection under the skin
* Treatment with exon skipping therapies 6 months prior to study start
* Treatment with ataluren or any investigational drug currently or within 5 half-lives prior to study start

Ages: 5 Years to 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2015-12-02 (Actual); Primary Completion 2018-02-08 (Actual); Study Completion 2020-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (12):
- United States (10):
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of Florida, Gainesville, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Saint Louis Children's Hospital, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
- Canada (2):
  - Alberta Children's Hospital, Calgary, Alberta
  - Children'S Hospital of Eastern Ontario, Ottawa, Ontario

REFERENCES:
- [Derived] Muntoni F, Byrne BJ, McMillan HJ, Ryan MM, Wong BL, Dukart J, Bansal A, Cosson V, Dreghici R, Guridi M, Rabbia M, Staunton H, Tirucherai GS, Yen K, Yuan X, Wagner KR; Taldefgrobep Alfa Study Group. The Clinical Development of Taldefgrobep Alfa: An Anti-Myostatin Adnectin for the Treatment of Duchenne Muscular Dystrophy. Neurol Ther. 2024 Feb;13(1):183-219. doi: 10.1007/s40120-023-00570-w. Epub 2024 Jan 8. PMID 38190001
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Doses for this study are based upon achieving a moderate to high degree of suppression in serum free myostatin at steady-state trough across 3 dose levels. A body weight-tiered, fixed-dose strategy targeting moderate (>50%), high (>85%) and near complete (>95%) suppression of serum free myostatin was used to select the three doses for the study.
Pre-assignment Details: Starting at Week 5, participants whose weight exceeded or dropped below the dosing weight tier to which they were assigned (by >1kg) were assigned to the new corresponding body weight-based dose within the participants assigned panel.
Groups:
- Panel 1 RO7239361: RO7239361 subcutaneous injections on specified days. The Panel 1 dose targets achievement of > 50% suppression in levels of free myostatin at trough after 5 weeks of weekly dosing. The Panel 1 body weight tier dose is >15kg at a dose of 4 mg (milligram) /0.8 mL (millilitre).
- Panel 2 RO7239361: RO7239361 subcutaneous injections on specified days. The Panel 2 dose targets achievement of > 85% suppression in levels of free myostatin at trough after 5 weeks of weekly dosing. Panel 2 body weight tier doses are =>15kg to =< 45kg at a dose of 12.5 mg /0.25 mL and =>45kg at a dose of 20 mg /0.4 mL
- Panel 3 and Expansion Panel RO7239361: RO7239361 subcutaneous injections on specified days. The Panel 3 and Expansion Panel dose targets achievement of > 95% suppression in levels of free myostatin at trough after 5 weeks of weekly dosing. Panel 3 and Expansion body weight tier doses are =>15kg to =< 45kg at a dose of 35 mg /0.7 mL and =>45kg at a dose of 50 mg /1.0 mL
Period: 24 Week Double-Blind Phase
Arm/Group | Placebo | Panel 1 RO7239361 | Panel 2 RO7239361 | Panel 3 and Expansion Panel RO7239361
Started | 11 | 7 | 6 | 19
Completed | 11 | 7 | 6 | 19
Not Completed | 0 | 0 | 0 | 0
Period: 228 Week Open-Label Phase
Arm/Group | Placebo | Panel 1 RO7239361 | Panel 2 RO7239361 | Panel 3 and Expansion Panel RO7239361
Started (Participants assigned to placebo in the double blind phase switched to RO for the open-label phase) | 0 (Double-blind (DB) placebo participants switched to RO7239361 (RO) for the open label phase.) | 9 (2 DB placebo participants switched to the Panel 1 RO cohort for the open-label phase.) | 8 (2 DB placebo participants switched to the Panel 2 RO cohort for the open-label phase.) | 26 (7 DB placebo participants switched to the Panel 3/Expansion RO cohort for the open-label phase.)
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 9 | 8 | 26
Not completed — Other | 0 | 0 | 1 | 4
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0
Not completed — Subject Request to Discontinue Treatment | 0 | 0 | 2 | 3
Not completed — Administrative Reason by Sponsor | 0 | 7 | 2 | 17
Not completed — Missing | 0 | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Doses tested in this study were based upon achieving and maintaining moderate (> 50% suppression), high (> 85%), and near complete (> 95%) suppression of serum free myostatin levels for Panels 1, 2, and 3 and Expansion Panel, respectively. Panel 3 was expanded after at least 2 weeks of dosing had been complete by at least 6 participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Panel 1 RO7239361 | Panel 2 RO7239361 | Panel 3 and Expansion Panel RO7239361 | Total
Number analyzed (Participants) | 11 | 7 | 6 | 19 | 43
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.8 (1.33) | 8.0 (2.24) | 8.0 (1.79) | 8.1 (1.81) | 8.2 (1.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 11 | 7 | 6 | 19 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2 | 4
  Not Hispanic or Latino | 9 | 7 | 5 | 13 | 34
  Unknown or Not Reported | 1 | 0 | 0 | 4 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 2 | 0 | 2 | 5 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1
  White | 9 | 6 | 3 | 13 | 31
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety Summary for the 24 Week Double-Blind Phase
Description: Percentage of participants with fatalities, adverse event (AEs) and serious adverse events (SAEs) up to Week 24.
  Participants in Panel 1 received 4 mg RO7239361; participants in Panel 2 received either 12.5 mg (weight between 15 and 45 kg) or 20 mg (weight >45 kg) RO7239361, and participants in Panel 3 and the Expansion Panel received either 35 mg (weight between 15 and 45 kg) or 50 mg (weight >45 kg) RO7239361.
Time Frame: Baseline to Week 24
Measure: Number; unit: percentage of participants
Groups:
- Panel 3 and Expansion RO7239361: RO7239361 subcutaneous injections on specified days. The Panel 3 and Expansion Panel dose targets achievement of > 95% suppression in levels of free myostatin at trough after 5 weeks of weekly dosing. Panel 3 and Expansion body weight tier doses are =>15kg to =< 45kg at a dose of 35 mg /0.7 mL and =>45kg at a dose of 50 mg /1.0 mL
Arm/Group | Placebo | Panel 1 RO7239361 | Panel 2 RO7239361 | Panel 3 and Expansion RO7239361
Number analyzed (Participants) | 11 | 7 | 6 | 19
percentage of participants
  Death | 0 | 0 | 0 | 0
  Adverse Events (AEs) | 81.8 | 71.4 | 100.0 | 94.7
  AEs leading to study withdrawal | 0 | 0 | 0 | 0
  Serious Adverse Events (SAE) | 9.1 | 0 | 0 | 5.3
  Very Severe AEs | 0 | 0 | 0 | 0
  Severe AEs | 0 | 0 | 0 | 0
  Related AEs | 27.3 | 14.3 | 50.0 | 36.8

2. Primary Outcome: Safety Summary up to Week 72
Description: Percentage of participants with fatalities, adverse event (AEs) and serious adverse events (SAEs) up to Week 72.
  Participants in Panel 1 received 4 mg RO7239361; participants in Panel 2 received either 12.5 mg (weight between 15 and 45 kg) or 20 mg (weight >45 kg) RO7239361, and participants in Panel 3 and the Expansion Panel received either 35 mg (weight between 15 and 45 kg) or 50 mg (weight >45 kg) RO7239361.
Time Frame: Baseline to Week 72
Measure: Number; unit: percentage of participants
Arm/Group | Panel 1 RO7239361 | Panel 2 RO7239361 | Panel 3 and Expansion Panel RO7239361
Number analyzed (Participants) | 9 | 8 | 26
percentage of participants
  Death | 0 | 0 | 0
  Adverse Events (AEs) | 100.0 | 100.0 | 96.2
  AEs leading to study withdrawal | 0 | 0 | 0
  Serious Adverse Events (SAE) | 0 | 25.0 | 7.7
  Very Severe AEs | 0 | 0 | 0
  Severe AEs | 0 | 25.0 | 3.8
  Related AEs | 77.8 | 62.5 | 50.0

3. Secondary Outcome: Maximum Observed Serum Concentrations (Cmax) of RO7239361 at Steady State for 4 mg QW, 12.5 mg QW and 35 mg QW Doses.
Description: PK parameter estimates at steady state. Steady state was achieved following approximately 12 weeks QW administration.
  Panel: 1 = 4mg QW, 2 = 12.5mg QW, 3 = 35mg QW
  Participants in Panel 1 received 4 mg RO7239361; participants in Panel 2 received either 12.5 mg (weight between 15 and 45 kg) or 20 mg (weight >45 kg) RO7239361, and participants in Panel 3 and the Expansion Panel received either 35 mg (weight between 15 and 45 kg) or 50 mg (weight >45 kg) RO7239361. No participants received the Panel 2 20mg dose.
Time Frame: Day 1: predose, 3, 6, 72 and 96 hours (h) postdose; Days 8, 15 and 22: predose; Day 29: predose and 96 h postdose; Weeks 12 and 24: predose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | Panel 1 RO7239361 | Panel 2 RO7239361 | Panel 3 and Expansion Panel RO7239361
Number analyzed (Participants) | 7 | 6 | 19
ng/ml | 3217 (15.8) | 8490 (21.5) | 24242 (26.3)

4. Secondary Outcome: Maximum Observed Serum Concentrations (Cmax) of RO7239361 at Steady State for 50 mg QW Dose.
Description: PK parameter estimates at steady state following approximately 12 weeks QW administration.
  Panel 3 = 50 mg QW
  Participants in Panel 1 received 4 mg RO7239361; participants in Panel 2 received either 12.5 mg (weight between 15 and 45 kg) or 20 mg (weight >45 kg) RO7239361, and participants in Panel 3 and the Expansion Panel received either 35 mg (weight between 15 and 45 kg) or 50 mg (weight >45 kg) RO7239361.
Time Frame: Day 1: predose, 3, 6, 72 and 96 h postdose; Days 8, 15 and 22: predose; Day 29: predose and 96 h postdose; Weeks 12 and 24: predose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Panel 3 and Expansion Panel RO7239361
Number analyzed (Participants) | 19
ng/mL | 23297 (NA) — Geometric Coefficient of Variation not evaluable as only one participant was included at this dose.

5. Secondary Outcome: Time of Maximum Observed Serum Concentrations (Tmax) of RO7239361 at Steady State for 4 mg QW, 12.5 mg QW and 35 mg QW Doses.
Description: PK parameter estimates at steady state. Steady state was achieved following approximately 12 weeks QW administration.
  Panel: 1 = 4mg QW, 2 = 12.5mg QW, 3 = 35mg QW.
  Results for the Panel 3 50mg QW dose level are represented in Outcome Measure 6. Participants in Panel 1 received 4 mg RO7239361; participants in Panel 2 received either 12.5 mg (weight between 15 and 45 kg) or 20 mg (weight >45 kg) RO7239361, and participants in Panel 3 and the Expansion Panel received either 35 mg (weight between 15 and 45 kg) or 50 mg (weight >45 kg) RO7239361.
Time Frame: as for outcome 4
Measure: Median (Full Range); unit: hour
Arm/Group | Panel 1 RO7239361 | Panel 2 RO7239361 | Panel 3 and Expansion Panel RO7239361
Number analyzed (Participants) | 7 | 6 | 18
hour | 28 [12 to 48] | 24 [11 to 47] | 30 [11 to 65]

6. Secondary Outcome: Time of Maximum Observed Serum Concentrations (Tmax) of RO7239361 at Steady State for 50 mg QW Dose.
Description: as for outcome 4
Time Frame: as for outcome 4
Measure: Median (Full Range); unit: hour
Arm/Group | Panel 3 and Expansion Panel RO7239361
Number analyzed (Participants) | 1
hour | 44 [NA to NA] — Geometric Coefficient of Variation not evaluable as only one participant was included at this dose.

7. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to Time of Next Dosing (AUCtau) of RO7239361 at Steady State for 4 mg QW, 12.5 mg QW and 35 mg QW Doses.
Description: PK parameter estimates at steady state. Steady state was achieved following approximately 12 weeks QW administration.
  Panel: 1 = 4mg QW, 2 = 12.5mg QW, 3 = 35mg QW
  Results for the Panel 3 50mg QW dose level are represented in Outcome Measure 8. Participants in Panel 1 received 4 mg RO7239361; participants in Panel 2 received either 12.5 mg (weight between 15 and 45 kg) or 20 mg (weight >45 kg) RO7239361, and participants in Panel 3 and the Expansion Panel received either 35 mg (weight between 15 and 45 kg) or 50 mg (weight >45 kg) RO7239361.
Time Frame: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•day/mL
Arm/Group | Panel 1 RO7239361 | Panel 2 RO7239361 | Panel 3 and Expansion Panel RO7239361
Number analyzed (Participants) | 7 | 6 | 18
ng•day/mL | 18676 (23) | 51461 (18) | 150609 (24)

8. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to Time of Next Dosing (AUCtau) of RO7239361 at Steady State for 50 mg QW Dose.
Description: as for outcome 4
Time Frame: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•day/mL
Arm/Group | Panel 3 and Expansion Panel RO7239361
Number analyzed (Participants) | 1
ng•day/mL | 151000 (NA) — Geometric Coefficient of Variation not evaluable as only one participant was included at this dose.

9. Secondary Outcome: RO7239361 Trough Concentrations
Description: Trough concentrations of RO7239361 at different dose levels.
  Panel 1 = 4mg, Panel 2 = 12.5mg and 20mg, Panel 3 = 35mg, Expansion Panels = 35mg and 50mg.
  Participants in Panel 1 received 4 mg RO7239361; participants in Panel 2 received either 12.5 mg (weight between 15 and 45 kg) or 20 mg (weight >45 kg) RO7239361, and participants in Panel 3 and the Expansion Panel received either 35 mg (weight between 15 and 45 kg) or 50 mg (weight >45 kg) RO7239361.
Time Frame: as for outcome 4
Population: Pharmacokinetic population. Panel 2, 20mg dose: the number of participants analyzed is 0 in those instances that the treatment was not administered at that visit.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Panel 2 RO7239361 12.5mg: RO7239361 subcutaneous injections on specified days. The Panel 2 dose targets achievement of > 85% suppression in levels of free myostatin at trough after 5 weeks of weekly dosing. Panel 2 body weight tier doses are =>15kg to =< 45kg at a dose of 12.5 mg /0.25 mL and =>45kg at a dose of 20 mg /0.4 mL
- Panel 2 RO7239361 20mg: RO7239361 subcutaneous injections on specified days. The Panel 2 dose targets achievement of > 85% suppression in levels of free myostatin at trough after 5 weeks of weekly dosing. Panel 2 body weight tier doses are =>15kg to =< 45kg at a dose of 12.5 mg /0.25 mL and =>45kg at a dose of 20 mg /0.4 mL.
  The dose was not administered at Days 1, 15, 22, 29 and 84.
- Panel 3 RO7239361 35mg: RO7239361 subcutaneous injections on specified days. RO7239361 subcutaneous injections on specified days, The Panel 2 dose targets achievement of > 85% suppression in levels of free myostatin at trough after 5 weeks of weekly dosing. Panel 2 body weight tier doses are =>15kg to =< 45kg at a dose of 12.5 mg /0.25 mL and =>45kg at a dose of 20 mg /0.4 mL
- Expansion Panel RO7239361 35mg; Expansion Panel RO7239361 50mg: RO7239361 subcutaneous injections on specified days. The Panel 3 and Expansion Panel dose targets achievement of > 95% suppression in levels of free myostatin at trough after 5 weeks of weekly dosing. Panel 3 and Expansion body weight tier doses are =>15kg to =< 45kg at a dose of 35 mg /0.7 mL and =>45kg at a dose of 50 mg /1.0 mL
Arm/Group | Panel 1 RO7239361 | Panel 2 RO7239361 12.5mg | Panel 2 RO7239361 20mg | Panel 3 RO7239361 35mg | Expansion Panel RO7239361 35mg | Expansion Panel RO7239361 50mg
Number analyzed (Participants) | 9 | 7 | 1 | 7 | 16 | 1
ng/mL
  Day 1: number analyzed (Participants) | 7 | 6 | 0 | 5 | 12 | 1
  Day 1 | 825.343 (23) | 2115.951 (20) |  | 6559.364 (26) | 6017.978 (23) | 5020.000 (NA) — Geometric Coefficient of Variation not evaluable as only one participant was included at this dose and therefore there was no dispersion.
  Day 15: number analyzed (Participants) | 7 | 6 | 0 | 6 | 12 | 1
  Day 15 | 1258.746 (35) | 3697.590 (20) |  | 9957.352 (34) | 9944.183 (24) | 9980.000 (NA) — Geometric Coefficient of Variation not evaluable as only one participant was included at this dose and therefore there was no dispersion.
  Day 22: number analyzed (Participants) | 5 | 6 | 0 | 5 | 11 | 1
  Day 22 | 1640.052 (15) | 4220.280 (32) |  | 12383.747 (30) | 13215.188 (24) | NA (NA) — Not evaluable, no sample taken
  Day 29: number analyzed (Participants) | 7 | 6 | 0 | 6 | 12 | 1
  Day 29 | 2015.695 (32) | 5107.668 (25) |  | 14110.005 (34) | 15094.455 (19) | NA (NA) — Not evaluable, no sample taken
  Day 84: number analyzed (Participants) | 8 | 6 | 0 | 7 | 16 | 1
  Day 84 | 2179.385 (26) | 6484.502 (19) |  | 19332.421 (20) | 18789.382 (18) | 27800.000 (NA) — Geometric Coefficient of Variation not evaluable as only one participant was included at this dose and therefore there was no dispersion.
  Day 168: number analyzed (Participants) | 9 | 7 | 1 | 7 | 14 | 1
  Day 168 | 2438.595 (16) | 6100.315 (25) | 6340.000 (NA) — Geometric Coefficient of Variation not evaluable as only one participant was included at this dose and therefore there was no dispersion. | 19923.182 (41) | 12580.299 (41) | 26200.000 (NA) — Geometric Coefficient of Variation not evaluable as only one participant was included at this dose and therefore there was no dispersion.

10. Secondary Outcome: Percentage of Participants With Positive Anti-RO7239361 Antibodies (ADA) Assessment, Double-Blind Phase
Description: A positive ADA sample is defined as one in which the presence of detectable ADAs is confirmed to be specific to RO7239361. A participant is considered as ADA positive if, after initiation of treatment, they have an ADA positive relative to baseline sample.
  Participants in Panel 1 received 4 mg RO7239361; participants in Panel 2 received either 12.5 mg (weight between 15 and 45 kg) or 20 mg (weight >45 kg) RO7239361, and participants in Panel 3 and the Expansion Panel received either 35 mg (weight between 15 and 45 kg) or 50 mg (weight >45 kg) RO7239361.
Time Frame: Day 8 through Week 24, baseline and on-study information represented in table.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Panel 1 RO7239361 | Panel 2 RO7239361 | Panel 3 and Expansion Panel RO7239361
Number analyzed (Participants) | 11 | 7 | 6 | 19
percentage of participants
  Baseline (BL): ADA Positive | 0 | 0 | 0 | 0
  BL: ADA Negative | 0 | 71.4 | 100.0 | 89.5
  BL: Missing | 100.0 | 28.6 | 0 | 10.5
  On-treatment: ADA Positive | 0 | 0 | 0 | 0
  On-treatment: Persistent Positive | 0 | 0 | 0 | 0
  On-treatment: Only last sample Positive | 0 | 0 | 0 | 0
  On-treatment: Other Positive | 0 | 0 | 0 | 0
  On-treatment: ADA Negative | 0 | 100.0 | 100.0 | 100.0
  On-treatment: ADA Negative, BL Positive, No Boost | 0 | 0 | 0 | 0
  On-treatment: Missing | 100.0 | 0 | 0 | 0

11. Secondary Outcome: Percentage of Participants With Positive Anti-RO7239361 Antibodies (ADA) Assessment up to Week 72
Description: A positive ADA sample is defined as one in which the presence of detectable ADAs is confirmed to be specific to RO7239361. A participant is considered as ADA positive if, after initiation of treatment, they have an ADA positive relative to baseline sample.
  Double-blind phase data for placebo participants is not included. Placebo participants in each arm moved on to RO7239361 upon entering the open label phase.
  Participants in Panel 1 received 4 mg RO7239361; participants in Panel 2 received either 12.5 mg (weight between 15 and 45 kg) or 20 mg (weight >45 kg) RO7239361, and participants in Panel 3 and the Expansion Panel received either 35 mg (weight between 15 and 45 kg) or 50 mg (weight >45 kg) RO7239361.
Time Frame: Day 8 through Week 72, baseline and on-study information represented in table.
Measure: Number; unit: percentage of participants
Arm/Group | Panel 1 RO7239361 | Panel 2 RO7239361 | Panel 3 and Expansion Panel RO7239361
Number analyzed (Participants) | 9 | 8 | 26
percentage of participants
  Baseline (BL): ADA Positive | 0 | 0 | 0
  BL: ADA Negative | 77.8 | 87.5 | 88.5
  BL: Missing | 22.2 | 12.5 | 11.5
  On-treatment: ADA Positive | 0 | 0 | 3.8
  On-treatment: Persistent Positive | 0 | 0 | 0
  On-treatment: Only last sample Positive | 0 | 0 | 3.8
  On-treatment: Other Positive | 0 | 0 | 0
  On-treatment: ADA Negative | 100.0 | 100.0 | 96.2
  On-treatment: ADA Negative, BL Positive, No Boost | 0 | 0 | 0
  On-treatment: Missing | 0 | 0 | 0

12. Secondary Outcome: Serum Concentration of Free Myostatin in the Double-Blind Phase
Description: Participants in Panel 1 received 4 mg RO7239361; participants in Panel 2 received either 12.5 mg (weight between 15 and 45 kg) or 20 mg (weight >45 kg) RO7239361, and participants in Panel 3 and the Expansion Panel received either 35 mg (weight between 15 and 45 kg) or 50 mg (weight >45 kg) RO7239361.
Time Frame: Baseline through Week 24
Population: The pharmacodynamics (PD) data set included all available data from subjects for whom PD measurements were available at baseline and at least one other timepoint.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | Panel 1 RO7239361 | Panel 2 RO7239361 | Panel 3 and Expansion Panel RO7239361
Number analyzed (Participants) | 11 | 7 | 6 | 19
pg/mL
  Baseline: number analyzed (Participants) | 11 | 6 | 6 | 16
  Baseline | 1405.1 (809.57) | 815.3 (155.14) | 1391.3 (1084.97) | 1121.8 (526.45)
  Day 4: number analyzed (Participants) | 8 | 5 | 4 | 18
  Day 4 | 1356.6 (641.27) | 421.4 (70.60) | 321.3 (165.91) | 58.3 (33.20)
  Day 5: number analyzed (Participants) | 9 | 7 | 6 | 18
  Day 5 | 1438.2 (809.18) | 446.6 (108.81) | 357.8 (166.27) | 66.1 (39.07)
  Day 8: number analyzed (Participants) | 10 | 6 | 6 | 19
  Day 8 | 1014.2 (549.26) | 522.7 (131.51) | 479.2 (319.13) | 206.8 (419.21)
  Day 15 | 1266.9 (611.27) | 478.4 (111.44) | 280.8 (148.53) | 54.8 (61.85)
  Day 22: number analyzed (Participants) | 11 | 7 | 6 | 17
  Day 22 | 1317.1 (728.48) | 382.4 (82.58) | 284.8 (324.16) | 35.3 (51.45)
  Day 29: number analyzed (Participants) | 11 | 7 | 6 | 17
  Day 29 | 1214.0 (676.80) | 372.3 (79.97) | 179.0 (137.39) | 24.8 (27.24)
  Day 33: number analyzed (Participants) | 11 | 7 | 6 | 18
  Day 33 | 1141.4 (606.99) | 291.1 (77.55) | 115.7 (84.49) | 24.3 (30.64)
  Week 12: number analyzed (Participants) | 10 | 6 | 4 | 18
  Week 12 | 1366.5 (631.28) | 307.8 (97.84) | 110.8 (49.80) | 16.2 (11.60)
  Week 24: number analyzed (Participants) | 11 | 7 | 6 | 18
  Week 24 | 1194.0 (599.59) | 297.1 (74.62) | 160.8 (122.75) | 23.4 (25.34)

13. Secondary Outcome: Percent Inhibition of Free Myostatin in the Double-Blind Phase
Description: as for outcome 12
Time Frame: Baseline through Week 24
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: percentage inhibition
Arm/Group | Placebo | Panel 1 RO7239361 | Panel 2 RO7239361 | Panel 3 and Expansion Panel RO7239361
Number analyzed (Participants) | 11 | 7 | 6 | 19
percentage inhibition
  Day 4: number analyzed (Participants) | 8 | 5 | 4 | 18
  Day 4 | 0.595 (23.6952) | 49.689 (11.7394) | 73.533 (9.8637) | 95.334 (2.4477)
  Day 5: number analyzed (Participants) | 9 | 7 | 6 | 18
  Day 5 | 3.114 (20.3395) | 46.506 (9.0917) | 69.700 (10.3411) | 94.545 (2.7608)
  Day 8: number analyzed (Participants) | 10 | 6 | 6 | 19
  Day 8 | 23.917 (31.1378) | 38.411 (7.0320) | 62.524 (9.7074) | 84.797 (22.1958)
  Day 15 | 5.744 (18.6190) | 40.763 (10.0071) | 77.090 (6.2939) | 96.488 (1.9665)
  Day 22: number analyzed (Participants) | 11 | 7 | 6 | 17
  Day 22 | 5.561 (11.7425) | 51.836 (9.3488) | 81.693 (5.7392) | 97.927 (1.1259)
  Day 29: number analyzed (Participants) | 11 | 7 | 6 | 17
  Day 29 | 12.599 (16.1591) | 52.926 (6.6001) | 86.894 (2.9590) | 98.202 (1.4590)
  Day 33: number analyzed (Participants) | 11 | 7 | 6 | 18
  Day 33 | 15.662 (17.3640) | 61.796 (4.5760) | 91.557 (2.6444) | 97.042 (5.4443)
  Week 12: number analyzed (Participants) | 10 | 6 | 4 | 18
  Week 12 | 5.289 (15.5082) | 60.254 (9.4283) | 92.454 (1.7243) | 98.415 (1.2882)
  Week 24: number analyzed (Participants) | 11 | 7 | 6 | 18
  Week 24 | 9.910 (17.8109) | 63.790 (5.7031) | 88.392 (5.1669) | 97.921 (2.2143)

14. Secondary Outcome: Serum Concentration of Drug-Myostatin Complex in the Double-Blind Phase
Description: as for outcome 12
Time Frame: Baseline through Week 24
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | Panel 1 RO7239361 | Panel 2 RO7239361 | Panel 3 and Expansion Panel RO7239361
Number analyzed (Participants) | 11 | 7 | 6 | 19
ng/mL
  Day 4: number analyzed (Participants) | 9 | 3 | 4 | 7
  Day 4 | 1.178 (1.8833) | 5.070 (0.9456) | 12.606 (5.7623) | 14.696 (5.7926)
  Day 5: number analyzed (Participants) | 8 | 5 | 6 | 6
  Day 5 | 2.119 (2.9826) | 5.845 (2.5725) | 14.856 (7.6131) | 17.308 (7.5955)
  Day 8: number analyzed (Participants) | 10 | 6 | 6 | 7
  Day 8 | 4.924 (12.9975) | 7.041 (2.3470) | 19.906 (9.8664) | 21.609 (11.0880)
  Day 15: number analyzed (Participants) | 11 | 7 | 6 | 7
  Day 15 | 0.613 (0.2102) | 14.067 (7.1096) | 29.229 (10.4929) | 45.289 (18.7600)
  Day 22: number analyzed (Participants) | 10 | 7 | 6 | 6
  Day 22 | 1.326 (1.3410) | 11.985 (4.8243) | 36.811 (26.8560) | 52.841 (21.5542)
  Day 29: number analyzed (Participants) | 11 | 7 | 6 | 7
  Day 29 | 1.593 (3.1007) | 15.735 (4.2010) | 43.236 (34.0300) | 67.255 (27.9376)
  Day 33: number analyzed (Participants) | 9 | 7 | 4 | 7
  Day 33 | 1.157 (1.0036) | 18.542 (3.9874) | 46.279 (24.1457) | 77.142 (32.4153)
  Week 12: number analyzed (Participants) | 10 | 6 | 5 | 14
  Week 12 | 7.082 (15.2289) | 28.556 (22.7890) | 79.555 (17.2126) | 88.402 (29.8080)
  Week 24: number analyzed (Participants) | 8 | 7 | 5 | 7
  Week 24 | 3.589 (7.8108) | 25.997 (6.4384) | 83.262 (64.2281) | 101.406 (45.4197)

15. Secondary Outcome: Fold Change From Baseline in Contractile Versus Non-contractile Content for Muscles in the Right Thigh in the Double-Blind Phase
Description: Ratio of contractile vs non-contractile content is contractile content / non-contractile content. Fold change from baseline of the ratio is defined as the ratio of fold change from baseline of contractile content vs fold change from baseline of non-contractile content.
  Right thigh measurements. W12 = Week 12, W24 = Week 24.
  Participants in Panel 1 received 4 mg RO7239361; participants in Panel 2 received either 12.5 mg (weight between 15 and 45 kg) or 20 mg (weight >45 kg) RO7239361, and participants in Panel 3 and the Expansion Panel received either 35 mg (weight between 15 and 45 kg) or 50 mg (weight >45 kg) RO7239361.
Time Frame: Baseline through Week 24
Population: The pharmacodynamics (PD) data set includes all available data from subjects for whom PD measurements are available at baseline and at least one other timepoint.
Measure: Mean (Standard Error); unit: Fold Change
Groups:
- Panel 3 RO7239361; Expansion Panel RO7239361: RO7239361 subcutaneous injections on specified days. The Panel 3 and Expansion Panel dose targets achievement of > 95% suppression in levels of free myostatin at trough after 5 weeks of weekly dosing. Panel 3 and Expansion body weight tier doses are =>15kg to =< 45kg at a dose of 35 mg /0.7 mL and =>45kg at a dose of 50 mg /1.0 mL
Arm/Group | Placebo | Panel 1 RO7239361 | Panel 2 RO7239361 | Panel 3 RO7239361 | Expansion Panel RO7239361
Number analyzed (Participants) | 11 | 7 | 6 | 6 | 13
Fold Change
  W12: ADDUCTOR LONGUS: number analyzed (Participants) | 7 | 3 | 5 | 4 | 11
  W12: ADDUCTOR LONGUS | 1.04 (0.291) | 0.95 (0.088) | 1.16 (0.330) | 2.27 (1.122) | 2.36 (0.875)
  W12: ADDUCTOR MAGNUS: number analyzed (Participants) | 8 | 5 | 4 | 5 | 11
  W12: ADDUCTOR MAGNUS | 0.69 (0.104) | 0.88 (0.283) | 1.12 (0.281) | 0.93 (0.255) | 1.04 (0.101)
  W12: BICEPS FEMORIS LONG: number analyzed (Participants) | 7 | 4 | 6 | 4 | 11
  W12: BICEPS FEMORIS LONG | 0.78 (0.221) | 0.94 (0.304) | 1.57 (0.556) | 1.10 (0.280) | 1.26 (0.237)
  W12: BICEPS FEMORIS SHORT: number analyzed (Participants) | 7 | 4 | 4 | 5 | 11
  W12: BICEPS FEMORIS SHORT | 0.92 (0.269) | 2.77 (1.144) | 2.03 (1.564) | 0.79 (0.162) | 1.31 (0.301)
  W12: GRACILIS: number analyzed (Participants) | 6 | 4 | 4 | 4 | 11
  W12: GRACILIS | 1.13 (0.318) | 7.57 (5.372) | 0.98 (0.176) | 3.41 (2.474) | 5.42 (3.871)
  W12:RECTUS FEMORIS: number analyzed (Participants) | 7 | 6 | 6 | 4 | 11
  W12:RECTUS FEMORIS | 0.74 (0.185) | 0.55 (0.134) | 4.49 (2.729) | 0.99 (0.345) | 2.02 (0.764)
  W12: SARTORIUS: number analyzed (Participants) | 6 | 4 | 5 | 4 | 10
  W12: SARTORIUS | 1.78 (0.771) | 0.69 (0.307) | 1.04 (0.443) | 0.90 (0.396) | 2.00 (0.683)
  W12: SEMIMEMBRANOSUS: number analyzed (Participants) | 8 | 5 | 6 | 6 | 13
  W12: SEMIMEMBRANOSUS | 0.82 (0.230) | 0.82 (0.284) | 1.47 (0.777) | 0.86 (0.276) | 1.31 (0.194)
  W12: SEMITENDINOSUS: number analyzed (Participants) | 8 | 4 | 5 | 4 | 11
  W12: SEMITENDINOSUS | 0.78 (0.262) | 2.95 (1.016) | 1.31 (0.260) | 1.42 (0.317) | 1.17 (0.160)
  W12: VASTUS INTERMEDIUS: number analyzed (Participants) | 7 | 3 | 4 | 4 | 10
  W12: VASTUS INTERMEDIUS | 2.59 (1.749) | 1.11 (0.292) | 0.62 (0.258) | 0.86 (0.157) | 1.64 (0.377)
  W12: VASTUS LATERALIS: number analyzed (Participants) | 7 | 5 | 6 | 5 | 12
  W12: VASTUS LATERALIS | 0.66 (0.160) | 0.89 (0.272) | 1.10 (0.333) | 1.78 (0.455) | 1.70 (0.334)
  W12: VASTUS MEDIALIS: number analyzed (Participants) | 6 | 4 | 6 | 4 | 12
  W12: VASTUS MEDIALIS | 1.08 (0.269) | 1.26 (0.112) | 2.97 (1.981) | 0.85 (0.280) | 5.96 (3.376)
  W24: ADDUCTOR LONGUS: number analyzed (Participants) | 9 | 4 | 4 | 5 | 11
  W24: ADDUCTOR LONGUS | 0.81 (0.290) | 1.14 (0.269) | 1.11 (0.471) | 1.36 (0.718) | 2.41 (0.813)
  W24: ADDUCTOR MAGNUS: number analyzed (Participants) | 10 | 6 | 4 | 5 | 11
  W24: ADDUCTOR MAGNUS | 0.66 (0.112) | 0.94 (0.296) | 0.59 (0.144) | 1.61 (0.697) | 1.14 (0.146)
  W24: BICEPS FEMORIS LONG: number analyzed (Participants) | 8 | 5 | 5 | 4 | 12
  W24: BICEPS FEMORIS LONG | 1.07 (0.511) | 1.13 (0.315) | 1.00 (0.349) | 1.29 (0.238) | 2.10 (1.044)
  W24: BICEPS FEMORIS SHORT: number analyzed (Participants) | 7 | 5 | 4 | 5 | 12
  W24: BICEPS FEMORIS SHORT | 0.91 (0.195) | 2.24 (1.027) | 2.15 (1.003) | 1.24 (0.411) | 2.02 (0.416)
  W24: GRACILIS: number analyzed (Participants) | 9 | 3 | 3 | 4 | 9
  W24: GRACILIS | 1.43 (0.686) | 3.03 (2.564) | 1.37 (0.465) | 1.45 (0.748) | 5.17 (3.540)
  W24:RECTUS FEMORIS: number analyzed (Participants) | 8 | 6 | 5 | 4 | 11
  W24:RECTUS FEMORIS | 0.94 (0.256) | 0.84 (0.220) | 7.43 (6.216) | 0.80 (0.262) | 3.01 (1.612)
  W24: SARTORIUS: number analyzed (Participants) | 7 | 5 | 4 | 4 | 10
  W24: SARTORIUS | 1.90 (0.872) | 0.73 (0.207) | 0.78 (0.375) | 3.24 (1.850) | 2.45 (0.842)
  W24: SEMIMEMBRANOSUS: number analyzed (Participants) | 10 | 6 | 5 | 4 | 12
  W24: SEMIMEMBRANOSUS | 0.66 (0.126) | 0.90 (0.361) | 0.72 (0.157) | 0.94 (0.250) | 1.39 (0.256)
  W24: SEMITENDINOSUS: number analyzed (Participants) | 9 | 5 | 4 | 6 | 11
  W24: SEMITENDINOSUS | 0.56 (0.119) | 1.59 (0.520) | 1.43 (0.524) | 1.04 (0.254) | 1.22 (0.221)
  W24: VASTUS INTERMEDIUS: number analyzed (Participants) | 7 | 4 | 3 | 4 | 10
  W24: VASTUS INTERMEDIUS | 0.95 (0.412) | 1.47 (0.446) | 0.63 (0.355) | 0.96 (0.095) | 1.47 (0.318)
  W24: VASTUS LATERALIS: number analyzed (Participants) | 10 | 5 | 5 | 4 | 12
  W24: VASTUS LATERALIS | 0.78 (0.159) | 1.88 (0.905) | 1.45 (0.596) | 1.43 (0.256) | 2.03 (0.484)
  W24: VASTUS MEDIALIS: number analyzed (Participants) | 8 | 5 | 4 | 4 | 12
  W24: VASTUS MEDIALIS | 2.14 (0.889) | 5.16 (3.580) | 6.01 (5.478) | 1.29 (0.474) | 3.50 (1.390)

16. Secondary Outcome: Change From Baseline in Thigh Muscle Maximal Cross Sectional Area (CSAmax) in the Double-Blind Phase
Description: Right thigh measurements. W12 = Week 12, W24 = Week 24.
  Participants in Panel 1 received 4 mg RO7239361; participants in Panel 2 received either 12.5 mg (weight between 15 and 45 kg) or 20 mg (weight >45 kg) RO7239361, and participants in Panel 3 and the Expansion Panel received either 35 mg (weight between 15 and 45 kg) or 50 mg (weight >45 kg) RO7239361.
Time Frame: Baseline through Week 24
Population: as for outcome 15
Measure: Mean (Standard Error); unit: Percentage Change
Groups:
- Panel 3RO7239361; Expansion Panel RO7239361: RO7239361 subcutaneous injections on specified days. The Panel 3 and Expansion Panel dose targets achievement of > 95% suppression in levels of free myostatin at trough after 5 weeks of weekly dosing. Panel 3 and Expansion body weight tier doses are =>15kg to =< 45kg at a dose of 35 mg /0.7 mL and =>45kg at a dose of 50 mg /1.0 mL
Arm/Group | Placebo | Panel 1 RO7239361 | Panel 2 RO7239361 | Panel 3RO7239361 | Expansion Panel RO7239361
Number analyzed (Participants) | 11 | 7 | 6 | 6 | 13
Percentage Change
  W12: ADDUCTOR LONGUS: number analyzed (Participants) | 9 | 6 | 6 | 6 | 12
  W12: ADDUCTOR LONGUS | 7.29 (16.559) | 8.31 (11.767) | 5.85 (11.074) | 14.61 (9.755) | 29.98 (8.530)
  W12: ADDUCTOR MAGNUS: number analyzed (Participants) | 9 | 6 | 6 | 6 | 12
  W12: ADDUCTOR MAGNUS | 31.01 (24.708) | 24.12 (11.804) | -3.73 (29.037) | 53.20 (25.328) | 4.01 (54.787)
  W12: BICEPS FEMORIS LONG: number analyzed (Participants) | 9 | 6 | 6 | 6 | 12
  W12: BICEPS FEMORIS LONG | 34.24 (18.328) | 33.43 (35.009) | 16.72 (17.806) | 19.22 (9.802) | 23.93 (11.289)
  W12: BICEPS FEMORIS SHORT: number analyzed (Participants) | 9 | 6 | 6 | 6 | 12
  W12: BICEPS FEMORIS SHORT | 14.10 (7.724) | 7.45 (11.592) | 2.69 (13.733) | 18.68 (7.479) | 9.84 (3.882)
  W12: GRACILIS: number analyzed (Participants) | 9 | 6 | 6 | 6 | 12
  W12: GRACILIS | 20.14 (15.489) | 43.00 (28.539) | 15.28 (8.693) | 27.02 (5.686) | 23.22 (5.440)
  W12:RECTUS FEMORIS: number analyzed (Participants) | 9 | 6 | 6 | 6 | 12
  W12:RECTUS FEMORIS | -7.86 (14.391) | 10.33 (11.927) | -3.56 (14.175) | 34.91 (6.037) | 16.01 (9.888)
  W12: SARTORIUS: number analyzed (Participants) | 9 | 6 | 6 | 6 | 12
  W12: SARTORIUS | 11.26 (6.584) | 6.59 (11.952) | -0.85 (6.383) | 10.81 (11.017) | 18.20 (5.519)
  W12: SEMIMEMBRANOSUS: number analyzed (Participants) | 9 | 6 | 6 | 6 | 12
  W12: SEMIMEMBRANOSUS | 39.11 (15.041) | 32.57 (19.133) | 16.56 (19.998) | 46.70 (16.480) | 31.01 (10.564)
  W12: SEMITENDINOSUS: number analyzed (Participants) | 9 | 6 | 6 | 6 | 12
  W12: SEMITENDINOSUS | 25.03 (9.409) | -1.24 (10.973) | 33.00 (26.730) | 36.69 (14.802) | 40.10 (10.180)
  W12: VASTUS INTERMEDIUS: number analyzed (Participants) | 9 | 6 | 6 | 6 | 12
  W12: VASTUS INTERMEDIUS | 10.47 (12.160) | 23.35 (12.704) | -52.03 (71.421) | -0.81 (19.353) | 10.44 (7.344)
  W12: VASTUS LATERALIS: number analyzed (Participants) | 9 | 6 | 6 | 6 | 12
  W12: VASTUS LATERALIS | 31.47 (39.343) | 38.32 (19.570) | 14.08 (27.902) | 57.86 (34.026) | 22.73 (15.138)
  W12: VASTUS MEDIALIS: number analyzed (Participants) | 9 | 6 | 6 | 6 | 12
  W12: VASTUS MEDIALIS | -17.89 (19.358) | 15.65 (8.463) | -11.60 (15.849) | 21.14 (9.746) | 17.89 (6.788)
  W24: ADDUCTOR LONGUS: number analyzed (Participants) | 11 | 7 | 5 | 6 | 12
  W24: ADDUCTOR LONGUS | 11.69 (15.626) | 23.41 (13.199) | 12.81 (16.393) | 17.15 (15.484) | 44.12 (13.323)
  W24: ADDUCTOR MAGNUS: number analyzed (Participants) | 11 | 7 | 5 | 6 | 12
  W24: ADDUCTOR MAGNUS | 34.17 (24.918) | 21.90 (12.345) | -6.71 (37.311) | 45.05 (27.520) | 4.41 (52.393)
  W24: BICEPS FEMORIS LONG: number analyzed (Participants) | 11 | 7 | 5 | 6 | 12
  W24: BICEPS FEMORIS LONG | 39.21 (19.760) | 42.84 (22.086) | -5.32 (29.140) | 33.70 (12.073) | 31.33 (13.370)
  W24: BICEPS FEMORIS SHORT: number analyzed (Participants) | 11 | 7 | 5 | 6 | 12
  W24: BICEPS FEMORIS SHORT | 20.09 (9.818) | 11.83 (13.013) | -0.44 (16.183) | 30.01 (13.494) | 18.60 (5.394)
  W24: GRACILIS: number analyzed (Participants) | 11 | 7 | 5 | 6 | 12
  W24: GRACILIS | 8.14 (7.148) | 18.72 (16.757) | 11.21 (5.461) | 48.95 (17.064) | 40.15 (8.382)
  W24:RECTUS FEMORIS: number analyzed (Participants) | 11 | 7 | 5 | 6 | 12
  W24:RECTUS FEMORIS | 8.97 (10.214) | 7.68 (13.082) | -10.01 (16.121) | 55.65 (27.535) | 38.40 (14.293)
  W24: SARTORIUS: number analyzed (Participants) | 11 | 7 | 5 | 6 | 12
  W24: SARTORIUS | 10.75 (7.136) | 0.81 (8.143) | -14.18 (9.481) | 16.63 (4.476) | 25.51 (6.404)
  W24: SEMIMEMBRANOSUS: number analyzed (Participants) | 11 | 7 | 5 | 6 | 12
  W24: SEMIMEMBRANOSUS | 45.83 (14.896) | 30.01 (18.631) | -11.48 (24.468) | 61.03 (25.524) | 49.49 (12.011)
  W24: SEMITENDINOSUS: number analyzed (Participants) | 11 | 7 | 5 | 6 | 12
  W24: SEMITENDINOSUS | 32.00 (16.102) | 36.17 (23.285) | 24.16 (23.403) | 73.68 (17.594) | 62.55 (11.073)
  W24: VASTUS INTERMEDIUS: number analyzed (Participants) | 11 | 7 | 5 | 6 | 12
  W24: VASTUS INTERMEDIUS | 14.86 (15.072) | 43.01 (11.506) | -68.05 (86.362) | 41.63 (34.926) | 22.55 (8.284)
  W24: VASTUS LATERALIS: number analyzed (Participants) | 11 | 7 | 5 | 6 | 12
  W24: VASTUS LATERALIS | 12.95 (35.465) | 47.79 (26.178) | 32.64 (30.136) | 45.41 (43.774) | 46.87 (20.919)
  W24: VASTUS MEDIALIS: number analyzed (Participants) | 11 | 7 | 5 | 6 | 12
  W24: VASTUS MEDIALIS | -9.09 (11.856) | 9.82 (6.965) | -13.74 (29.664) | 10.46 (12.093) | 23.94 (11.321)

17. Secondary Outcome: Percentage of Participants With Positive Anti-RO7239361 Antibodies (ADA) Assessment, Whole Study
Description: A positive ADA sample is defined as one in which the presence of detectable ADAs is confirmed to be specific to RO7239361. A participant is considered as ADA positive if, after initiation of treatment, they have an ADA positive relative to baseline sample.
  Double-blind phase data for placebo participants are not included in this Whole Study outcome measure, but are reported in the outcome measure specific to the double-blind period. At the end of the double-blind period participants in the placebo arm switched to one of the RO7239361 arms upon entering the open label phase.
  Participants in Panel 1 received 4 mg RO7239361; participants in Panel 2 received either 12.5 mg (weight between 15 and 45 kg) or 20 mg (weight >45 kg) RO7239361, and participants in Panel 3 and the Expansion Panel received either 35 mg (weight between 15 and 45 kg) or 50 mg (weight >45 kg) RO7239361.
Time Frame: Day 8 through Week 228, baseline and on-study information represented in table.
Population: The safety population included all participants who received at least one dose of study drug. The Whole Study set reported here includes data from RO7239361-treated participants only.
Measure: Number; unit: percentage of participants
Arm/Group | Panel 1 RO7239361 | Panel 2 RO7239361 | Panel 3 and Expansion Panel RO7239361
Number analyzed (Participants) | 9 | 8 | 26
percentage of participants
  Baseline (BL): ADA Positive | 0 | 0 | 0
  BL: ADA Negative | 100.0 | 87.5 | 92.3
  BL: Missing | 0 | 12.5 | 7.7
  On-treatment: ADA Positive | 0 | 0 | 3.8
  On-treatment: Persistent Positive | 0 | 0 | 0
  On-treatment: Only last sample Positive | 0 | 0 | 0
  On-treatment: Other Positive | 0 | 0 | 3.8
  On-treatment: ADA Negative | 100.0 | 100.0 | 96.2
  On-treatment: ADA Negative, BL Positive, No Boost | 0 | 0 | 0
  On-treatment: Missing | 0 | 0 | 0

18. Secondary Outcome: Serum Concentration of Free Myostatin, Whole Study
Description: Double-blind phase data for placebo participants are not included in this Whole Study outcome measure, but are reported in the outcome measure specific to the double-blind period. At the end of the double-blind period participants in the placebo arm switched to one of the RO7239361 arms upon entering the open label phase.
  Participants in Panel 1 received 4 mg RO7239361; participants in Panel 2 received either 12.5 mg (weight between 15 and 45 kg) or 20 mg (weight >45 kg) RO7239361, and participants in Panel 3 and the Expansion Panel received either 35 mg (weight between 15 and 45 kg) or 50 mg (weight >45 kg) RO7239361.
Time Frame: Baseline through Week 252
Population: The pharmacodynamics (PD) data set included all available data from subjects for whom PD measurements were available at baseline and at least one other timepoint. The Whole Study set reported here includes data from RO7239361-treated participants only.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Panel 1 RO7239361 | Panel 2 RO7239361 | Panel 3 and Expansion Panel RO7239361
Number analyzed (Participants) | 9 | 8 | 25
pg/mL
  Baseline: number analyzed (Participants) | 8 | 8 | 23
  Baseline | 986.8 (363.69) | 1358.4 (964.47) | 1159.3 (601.29)
  Day 4: number analyzed (Participants) | 5 | 4 | 18
  Day 4 | 421.4 (70.60) | 321.3 (165.91) | 58.3 (33.20)
  Day 5: number analyzed (Participants) | 7 | 6 | 18
  Day 5 | 446.6 (108.81) | 357.8 (166.27) | 66.1 (39.07)
  Day 8: number analyzed (Participants) | 6 | 6 | 19
  Day 8 | 522.7 (131.51) | 479.2 (319.13) | 206.8 (419.21)
  Day 15: number analyzed (Participants) | 7 | 6 | 19
  Day 15 | 478.4 (111.44) | 280.8 (148.53) | 54.8 (61.85)
  Day 22: number analyzed (Participants) | 7 | 6 | 17
  Day 22 | 382.4 (82.58) | 284.8 (324.16) | 35.3 (51.45)
  Day 29: number analyzed (Participants) | 7 | 6 | 17
  Day 29 | 372.3 (79.97) | 179.0 (137.39) | 24.8 (27.24)
  Day 33: number analyzed (Participants) | 7 | 6 | 18
  Day 33 | 291.1 (77.55) | 115.7 (84.49) | 24.3 (30.64)
  Week 12: number analyzed (Participants) | 8 | 6 | 25
  Week 12 | 394.0 (179.78) | 115.0 (62.23) | 18.1 (13.37)
  Week 24: number analyzed (Participants) | 9 | 8 | 24
  Week 24 | 357.9 (137.56) | 139.1 (111.63) | 23.0 (23.68)
  Week 25: number analyzed (Participants) | 6 | 6 | 17
  Week 25 | 331.0 (116.78) | 154.5 (115.21) | 22.8 (18.48)
  Week 36: number analyzed (Participants) | 9 | 7 | 16
  Week 36 | 340.3 (98.24) | 81.4 (36.00) | 21.1 (22.03)
  Week 48: number analyzed (Participants) | 9 | 7 | 16
  Week 48 | 401.3 (233.76) | 79.0 (37.85) | 18.6 (12.11)
  Week 60: number analyzed (Participants) | 7 | 5 | 9
  Week 60 | 284.6 (96.92) | 90.4 (39.30) | 36.3 (54.13)
  Week 72: number analyzed (Participants) | 5 | 4 | 3
  Week 72 | 326.8 (151.29) | 132.0 (146.37) | 205.7 (321.58)
  Week 84: number analyzed (Participants) | 4 | 2 | 15
  Week 84 | 534.0 (260.31) | 74.2 (13.58) | 115.6 (146.44)
  Week 108: number analyzed (Participants) | 9 | 5 | 16
  Week 108 | 320.9 (222.10) | 84.4 (61.19) | 40.2 (42.70)
  Week 132: number analyzed (Participants) | 8 | 7 | 21
  Week 132 | 283.5 (103.73) | 71.0 (40.02) | 40.2 (38.26)
  Week 144: number analyzed (Participants) | 0 | 1 | 0
  Week 144 |  | 95.2 (NA) — NA: SD not calculable for 1 participant |
  Week 156: number analyzed (Participants) | 7 | 4 | 8
  Week 156 | 208.7 (64.52) | 48.9 (22.42) | 20.0 (0.00)
  Week 180: number analyzed (Participants) | 2 | 0 | 0
  Week 180 | 212.5 (146.37) |  |
  Week 252: number analyzed (Participants) | 0 | 1 | 0
  Week 252 |  | 20.0 (NA) — NA: SD not calculable for 1 participant |

19. Secondary Outcome: Percent Inhibition of Free Myostatin, Whole Study
Description: as for outcome 18
Time Frame: Baseline through Week 252
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: percentage inhibition
Arm/Group | Panel 1 RO7239361 | Panel 2 RO7239361 | Panel 3 and Expansion Panel RO7239361
Number analyzed (Participants) | 8 | 8 | 22
percentage inhibition
  Day 4: number analyzed (Participants) | 4 | 4 | 15
  Day 4 | 49.689 (11.7394) | 73.533 (9.8637) | 95.334 (2.4477)
  Day 5: number analyzed (Participants) | 6 | 6 | 16
  Day 5 | 46.506 (9.0917) | 69.700 (10.3411) | 94.545 (2.7608)
  Day 8: number analyzed (Participants) | 5 | 6 | 16
  Day 8 | 38.411 (7.0320) | 62.524 (9.7074) | 84.797 (22.1958)
  Day 15: number analyzed (Participants) | 6 | 6 | 16
  Day 15 | 40.763 (10.0071) | 77.090 (6.2939) | 96.488 (1.9665)
  Day 22: number analyzed (Participants) | 6 | 6 | 15
  Day 22 | 51.836 (9.3488) | 81.693 (5.7392) | 97.927 (1.1259)
  Day 29: number analyzed (Participants) | 6 | 6 | 15
  Day 29 | 52.926 (6.6001) | 86.894 (2.9590) | 98.202 (1.4590)
  Day 33: number analyzed (Participants) | 6 | 6 | 15
  Day 33 | 61.796 (4.5760) | 91.557 (2.6444) | 97.042 (5.4443)
  Week 12: number analyzed (Participants) | 7 | 6 | 22
  Week 12 | 58.934 (8.7345) | 92.025 (2.0548) | 98.208 (1.5605)
  Week 24: number analyzed (Participants) | 8 | 8 | 21
  Week 24 | 63.199 (5.3419) | 89.664 (5.0245) | 98.009 (1.8677)
  Week 25: number analyzed (Participants) | 5 | 6 | 16
  Week 25 | 62.446 (7.0668) | 88.689 (4.8868) | 97.974 (1.8259)
  Week 36: number analyzed (Participants) | 8 | 7 | 15
  Week 36 | 64.103 (5.3774) | 92.057 (2.6300) | 98.470 (0.8410)
  Week 48: number analyzed (Participants) | 8 | 7 | 14
  Week 48 | 58.161 (15.7101) | 92.237 (3.4952) | 98.036 (1.4516)
  Week 60: number analyzed (Participants) | 6 | 5 | 7
  Week 60 | 66.280 (8.4684) | 90.974 (2.1780) | 97.177 (2.8783)
  Week 72: number analyzed (Participants) | 4 | 4 | 3
  Week 72 | 65.956 (8.2066) | 92.536 (2.4445) | 79.193 (31.9504)
  Week 84: number analyzed (Participants) | 4 | 2 | 13
  Week 84 | 54.990 (11.0397) | 92.328 (5.7945) | 89.744 (13.0990)
  Week 108: number analyzed (Participants) | 8 | 5 | 14
  Week 108 | 70.498 (15.2905) | 92.412 (3.3662) | 95.884 (3.5214)
  Week 132: number analyzed (Participants) | 8 | 7 | 18
  Week 132 | 71.129 (4.9576) | 92.935 (3.8121) | 96.713 (2.4278)
  Week 144: number analyzed (Participants) | 0 | 1 | 0
  Week 144 |  | 94.732 (NA) — NA: SD not calculable for 1 participant |
  Week 156: number analyzed (Participants) | 6 | 4 | 6
  Week 156 | 74.712 (5.7764) | 94.881 (1.3726) | 98.183 (0.8086)
  Week 180: number analyzed (Participants) | 2 | 0 | 0
  Week 180 | 75.374 (9.5968) |  |
  Week 252: number analyzed (Participants) | 0 | 1 | 0
  Week 252 |  | 96.283 (NA) — NA: SD not calculable for 1 participant |

20. Secondary Outcome: Serum Concentration of Drug-Myostatin Complex, Whole Study
Description: Participants in the Placebo arm received placebo during the double-blind (DB) period (up to Week 24) and received RO7239361 during the open label (OL) phase. PFS in table row title indicates when study drug was changed from vial to prefilled syringe (PFS).
  Participants in Panel 1 received 4 mg RO7239361; participants in Panel 2 received either 12.5 mg (weight between 15 and 45 kg) or 20 mg (weight >45 kg) RO7239361, and participants in Panel 3 and the Expansion Panel received either 35 mg (weight between 15 and 45 kg) or 50 mg (weight >45 kg) RO7239361.
Time Frame: Baseline through Week 252
Population: The pharmacodynamics (PD) data set included all available data from subjects for whom PD measurements were available at baseline and at least one other timepoint. Data are analyzed according to the arms in which participants started the study.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Placebo, Then RO7239361: Placebo subcutaneous injections on specified days. At the end of the DB period these participants switched to treatment to treatment with RO7239361 at dose levels of either Panel 1, Panel 2 or Panel 3.
- Panel 1 RO7239361 Whole Study: RO7239361 subcutaneous injections on specified days. The Panel 1 dose targets achievement of > 50% suppression in levels of free myostatin at trough after 5 weeks of weekly dosing. The Panel 1 body weight tier dose is >15kg at a dose of 4 mg (milligram) /0.8 mL (millilitre).
- Panel 2 RO7239361 Whole Study: RO7239361 subcutaneous injections on specified days. The Panel 2 dose targets achievement of > 85% suppression in levels of free myostatin at trough after 5 weeks of weekly dosing. Panel 2 body weight tier doses are =>15kg to =< 45kg at a dose of 12.5 mg /0.25 mL and =>45kg at a dose of 20 mg /0.4 mL
- Panel 3 and Expansion Panel RO7239361 Whole Study: RO7239361 subcutaneous injections on specified days. The Panel 3 and Expansion Panel dose targets achievement of > 95% suppression in levels of free myostatin at trough after 5 weeks of weekly dosing. Panel 3 and Expansion body weight tier doses are =>15kg to =< 45kg at a dose of 35 mg /0.7 mL and =>45kg at a dose of 50 mg /1.0 mL
Arm/Group | Placebo, Then RO7239361 | Panel 1 RO7239361 Whole Study | Panel 2 RO7239361 Whole Study | Panel 3 and Expansion Panel RO7239361 Whole Study
Number analyzed (Participants) | 11 | 7 | 6 | 19
ng/mL
  Day 4: number analyzed (Participants) | 9 | 3 | 4 | 7
  Day 4 | 1.178 (1.8833) | 5.070 (0.9456) | 12.606 (5.7623) | 14.696 (5.7926)
  Day 5: number analyzed (Participants) | 8 | 5 | 6 | 6
  Day 5 | 2.119 (2.9826) | 5.845 (2.5725) | 14.856 (7.6131) | 17.308 (7.5955)
  Day 8: number analyzed (Participants) | 10 | 6 | 6 | 7
  Day 8 | 4.924 (12.9975) | 7.041 (2.3470) | 19.906 (9.8664) | 21.609 (11.0880)
  Day 15: number analyzed (Participants) | 11 | 7 | 6 | 7
  Day 15 | 0.613 (0.2102) | 14.067 (7.1096) | 29.229 (10.4929) | 45.289 (18.7600)
  Day 22: number analyzed (Participants) | 10 | 7 | 6 | 6
  Day 22 | 1.326 (1.3410) | 11.985 (4.8243) | 36.811 (26.8560) | 52.841 (21.5542)
  Day 29: number analyzed (Participants) | 11 | 7 | 6 | 7
  Day 29 | 1.593 (3.1007) | 15.735 (4.2010) | 43.236 (34.0300) | 67.255 (27.9376)
  Day 33: number analyzed (Participants) | 9 | 7 | 4 | 7
  Day 33 | 1.157 (1.0036) | 18.542 (3.9874) | 46.279 (24.1457) | 77.142 (32.4153)
  Week 12: number analyzed (Participants) | 10 | 6 | 5 | 14
  Week 12 | 7.082 (15.2289) | 28.556 (22.7890) | 79.555 (17.2126) | 88.402 (29.8080)
  Week 24 (end of DB period): number analyzed (Participants) | 8 | 7 | 5 | 7
  Week 24 (end of DB period) | 3.589 (7.8108) | 25.997 (6.4384) | 83.262 (64.2281) | 101.406 (45.4197)
  Week 25 (Week 1 OL): number analyzed (Participants) | 7 | 7 | 5 | 8
  Week 25 (Week 1 OL) | 3.186 (6.9734) | 31.963 (8.0240) | 77.926 (56.9987) | 102.211 (40.2284)
  Week 36 (Week 12 OL): number analyzed (Participants) | 10 | 6 | 5 | 14
  Week 36 (Week 12 OL) | 95.788 (88.1521) | 22.584 (8.6839) | 57.164 (25.8284) | 101.234 (42.0902)
  Week 48 (Week 24 OL): number analyzed (Participants) | 9 | 7 | 0 | 18
  Week 48 (Week 24 OL) | 90.593 (73.7102) | 27.461 (7.2306) |  | 103.657 (45.8802)
  Week 60 (Week 36 OL): number analyzed (Participants) | 5 | 7 | 5 | 3
  Week 60 (Week 36 OL) | 63.358 (37.5591) | 41.779 (34.2407) | 89.712 (38.9214) | 67.163 (8.4904)
  Week 72 (Week 48 OL): number analyzed (Participants) | 5 | 5 | 1 | 4
  Week 72 (Week 48 OL) | 92.086 (68.5222) | 26.740 (3.0256) | 0.550 (NA) — NA: SD not calculable for 1 participant | 102.025 (31.4717)
  Week 84 (Week 60 OL): number analyzed (Participants) | 6 | 2 | 0 | 16
  Week 84 (Week 60 OL) | 146.950 (131.3706) | 27.110 (3.2527) |  | 117.719 (41.1143)
  Week 108 (Week 84 OL): number analyzed (Participants) | 10 | 7 | 5 | 18
  Week 108 (Week 84 OL) | 122.610 (87.1911) | 36.014 (10.9338) | 66.020 (7.2878) | 114.806 (32.7432)
  Week 132 (Week 108 OL): number analyzed (Participants) | 9 | 6 | 5 | 18
  Week 132 (Week 108 OL) | 95.811 (48.1440) | 32.133 (8.2848) | 75.040 (14.3015) | 107.378 (37.8814)
  Week 144 (Week 120 OL): number analyzed (Participants) | 0 | 1 | 0 | 0
  Week 144 (Week 120 OL) |  | 25.600 (NA) — NA: SD not calculable for 1 participant |  |
  Week 156 (Week 132 OL): number analyzed (Participants) | 7 | 7 | 4 | 18
  Week 156 (Week 132 OL) | 95.529 (48.0065) | 30.186 (7.0053) | 69.325 (17.7064) | 108.100 (35.5833)
  Week 156 (Week 132 OL: Day 1 PFS): number analyzed (Participants) | 2 | 0 | 0 | 0
  Week 156 (Week 132 OL: Day 1 PFS) | 64.400 (0.5657) |  |  |
  Week 156 (Week 132 OL: Week 12 PFS): number analyzed (Participants) | 1 | 0 | 0 | 6
  Week 156 (Week 132 OL: Week 12 PFS) | 152.000 (NA) — NA: SD not calculable for 1 participant |  |  | 125.583 (44.4144)
  Week 168 (Week 144 OL: Day 1 PFS): number analyzed (Participants) | 3 | 0 | 3 | 3
  Week 168 (Week 144 OL: Day 1 PFS) | 105.700 (54.5772) |  | 70.100 (25.1213) | 122.633 (91.2542)
  Week 168 (Week 144 OL: Day 8 PFS): number analyzed (Participants) | 0 | 0 | 0 | 1
  Week 168 (Week 144 OL: Day 8 PFS) |  |  |  | 119.000 (NA) — NA: SD not calculable for 1 participant
  Week 168 (Week 144 OL: Week 12 PFS): number analyzed (Participants) | 0 | 0 | 1 | 0
  Week 168 (Week 144 OL: Week 12 PFS) |  |  | 94.900 (NA) — NA: SD not calculable for 1 participant |
  Week 180 (Week 156 OL): number analyzed (Participants) | 3 | 7 | 2 | 0
  Week 180 (Week 156 OL) | 45.933 (28.3161) | 25.589 (12.2478) | 103.300 (16.5463) |
  Week 180 (Week 156 OL: Week 12 PFS): number analyzed (Participants) | 0 | 1 | 0 | 0
  Week 180 (Week 156 OL: Week 12 PFS) |  | 62.600 (NA) — NA: SD not calculable for 1 participant |  |
  Week 192 (Week 168 OL: Day 1 PFS): number analyzed (Participants) | 0 | 1 | 0 | 0
  Week 192 (Week 168 OL: Day 1 PFS) |  | 18.000 (NA) — NA: SD not calculable for 1 participant |  |
  Week 192 (Week 168 OL: Day 45 PFS): number analyzed (Participants) | 0 | 1 | 0 | 0
  Week 192 (Week 168 OL: Day 45 PFS) |  | 80.400 (NA) — NA: SD not calculable for 1 participant |  |
  Week 252 (Week 228 OL): number analyzed (Participants) | 10 | 5 | 3 | 17
  Week 252 (Week 228 OL) | 96.770 (61.6084) | 52.680 (20.8619) | 87.900 (38.5763) | 106.071 (48.6434)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 252
Description: Upon completion of the double-blind phase, participants who were receiving placebo switched to the equivalent RO7239361 panel dose for the open label phase. All adverse event data is represented according to the phase (double-blind or open-label) during which the participant experienced the event.
Groups:
- Placebo Double-Blind: Placebo subcutaneous injections on specified days during the double-blind period.
- Panel 1 RO7239361 Double-Blind; Panel 2 RO7239361 Double-Blind; Panel 3 and Expansion Panel RO7239361 Double-Blind: RO7239361 subcutaneous injections on specified days during the double-blind period.
- Panel 1 RO7239361 Open-Label; Panel 3 and Expansion Panel RO7239361 Open-Label: RO7239361 subcutaneous injections on specified days during the open-label period.
- Panel 2 RO7239361 Open-Label: RO7239361 subcutaneous injections on specified days during the open label period.
Arm/Group | Placebo Double-Blind | Panel 1 RO7239361 Double-Blind | Panel 2 RO7239361 Double-Blind | Panel 3 and Expansion Panel RO7239361 Double-Blind | Panel 1 RO7239361 Open-Label | Panel 2 RO7239361 Open-Label | Panel 3 and Expansion Panel RO7239361 Open-Label
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/7 | 0/6 | 0/19 | 0/9 | 0/8 | 0/26
Serious Adverse Events (participants affected / at risk) | 1/11 | 0/7 | 0/6 | 1/19 | 1/9 | 2/8 | 1/26
Other Adverse Events (participants affected / at risk) | 9/11 | 5/7 | 6/6 | 17/19 | 9/9 | 6/8 | 24/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Double-Blind (N=11) | Panel 1 RO7239361 Double-Blind (N=7) | Panel 2 RO7239361 Double-Blind (N=6) | Panel 3 and Expansion Panel RO7239361 Double-Blind (N=19) | Panel 1 RO7239361 Open-Label (N=9) | Panel 2 RO7239361 Open-Label (N=8) | Panel 3 and Expansion Panel RO7239361 Open-Label (N=26)
APPENDICITIS PERFORATED (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SKULL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
CONVERSION DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Double-Blind (N=11) | Panel 1 RO7239361 Double-Blind (N=7) | Panel 2 RO7239361 Double-Blind (N=6) | Panel 3 and Expansion Panel RO7239361 Double-Blind (N=19) | Panel 1 RO7239361 Open-Label (N=9) | Panel 2 RO7239361 Open-Label (N=8) | Panel 3 and Expansion Panel RO7239361 Open-Label (N=26)
CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MYOCARDIAL FIBROSIS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SINUS TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DERMOID CYST (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
EAR PAIN (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TYMPANIC MEMBRANE HYPERAEMIA (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TYMPANIC MEMBRANE PERFORATION (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CUSHINGOID (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
DELAYED PUBERTY (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CATARACT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DRY EYE (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VISION BLURRED (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (11)
BREATH ODOUR (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 2 (4) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (3) | 9 (14)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTRIC ULCER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
LIP SWELLING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MALPOSITIONED TEETH (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MOUTH ULCERATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUCOUS STOOLS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 4 (11) | 1 (1) | 8 (9)
CHILLS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INJECTION SITE BRUISING (General disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 6 (13)
INJECTION SITE DISCOMFORT (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INJECTION SITE ERYTHEMA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 4 (6) | 0 (0) | 8 (13)
INJECTION SITE HAEMORRHAGE (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
INJECTION SITE IRRITATION (General disorders) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 5 (23) | 0 (0) | 0 (0)
INJECTION SITE OEDEMA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
INJECTION SITE PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 1 (1) | 2 (3)
INJECTION SITE PRURITUS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INJECTION SITE RASH (General disorders) | 1 (1) | 1 (1) | 1 (9) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
INJECTION SITE REACTION (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
INJECTION SITE SWELLING (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PERIPHERAL SWELLING (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 3 (3) | 0 (0) | 1 (1) | 5 (6) | 1 (1) | 2 (2) | 4 (8)
SEASONAL ALLERGY (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
ABSCESS ORAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BODY TINEA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CONJUNCTIVITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EAR INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 4 (5)
FUNGAL SKIN INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (5)
LABYRINTHITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NAIL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 1 (2) | 1 (1) | 4 (4) | 4 (7) | 1 (2) | 7 (12)
ONYCHOMYCOSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (4)
PNEUMONIA MYCOPLASMAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SCARLET FEVER (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
SKIN CANDIDA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
STAPHYLOCOCCAL SKIN INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TOOTH ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (3) | 0 (0) | 2 (2) | 4 (5) | 0 (0) | 1 (1) | 11 (25)
VIRAL RHINITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 4 (4)
CORNEAL ABRASION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EYE CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
EYELID CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 7 (20) | 0 (0) | 6 (8)
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
HEAD INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
JOINT INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
LIMB INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
POST-TRAUMATIC PAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SKIN ABRASION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SOFT TISSUE INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
SUNBURN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
THERMAL BURN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LYMPH NODE PALPABLE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 3 (4)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 5 (5)
COCCYDYNIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INTERVERTEBRAL DISC COMPRESSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
JOINT CONTRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
MUSCLE TIGHTNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 4 (4)
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1) | 7 (19) | 2 (3) | 0 (0) | 9 (27)
MOTOR DYSFUNCTION (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SINUS HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ANGER (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BRUXISM (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ENURESIS (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
POLYURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TESTICULAR TORSION (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 4 (5) | 7 (11)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (13)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LOWER RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 5 (5)
NASAL DISCHARGE DISCOLOURATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 4 (6)
PARANASAL SINUS HYPERSECRETION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (5)
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACNE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COLD SWEAT (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
EPHELIDES (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LIVEDO RETICULARIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (4) | 1 (2) | 0 (0) | 0 (0) | 2 (3)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FLUSHING (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HAEMATOMA (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-14): https://cdn.clinicaltrials.gov/large-docs/69/NCT02515669/Prot_SAP_000.pdf